CLINICAL TRIAL: NCT01769326
Title: Influence of Timing on Motor Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Steven C. Cramer, MD, Professor of Neurology, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS# 2008-6432; R43HD074331-01 (NIH)
Record Dates: First submitted 2012-11-16; First posted 2013-01-16 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MusicGlove Group (Experimental): Subject participates in 3 weeks of exercising with the experimental device: MusicGlove at a minimum of 3 days per week, 1 hour per day with the exercise program
  Interventions: Device: MusicGlove
- Control Group for Music Glove (Active Comparator): Subject participates in 3 weeks of conventional hand exercise program, at a minimum of 3 days per week, 1 hour per day with the exercise program.
  Interventions: Other: Conventional hand exercise
- Resonating Arm Exerciser (RAE) (Experimental): Subject participates in 3 weeks of exercising with the experimental device: RAE at a minimum of 3 days per week, 1 hour per day with the exercise program
  Interventions: Device: Resonating Arm Exerciser
- Control Group for RAE (Active Comparator): Subject participates in 3 weeks of conventional arm exercise program, at a minimum of 3 days per week, 1 hour per day with the exercise program.
  Interventions: Other: Conventional Arm Exercise

INTERVENTIONS:
Other: Conventional hand exercise — Conventional hand exercise consists of passive and active range of motion exercise, and simple coordination exercises with the fingers
  Arms: Control Group for Music Glove
Device: MusicGlove — The MusicGlove is a glove that detects different grip types. Subjects play a musical game by completing different grips.
  Arms: MusicGlove Group
Other: Conventional Arm Exercise — Conventional arm exercise consists of passive and active range of motion exercise, and simple weight bearing exercises
  Arms: Control Group for RAE
Device: Resonating Arm Exerciser — The RAE is a lever that attaches to a manual wheelchair with elastic bands and can be pushed back and forth to exercise the arm.
  Other Names: RAE
  Arms: Resonating Arm Exerciser (RAE)

SUMMARY:
The purpose of this research study is to compare different methods for training hand movement at home after stroke. This study involves research because it will test two experimental devices, the MusicGlove and the Resonating Arm Exerciser (RAE), compared to conventional hand and arm exercises. The MusicGlove is a glove that measures finger movements and allows its user to play a musical computer game using those movements. The RAE is a lever that attaches to a manual wheelchair with elastic bands and can be pushed back and forth to exercise the arm.

DETAILED DESCRIPTION:
The purpose of this research study is to compare different methods for training hand movement at home after stroke. This study involves research because it will test two experimental devices, the MusicGlove and the Resonating Arm Exerciser (RAE), compared to conventional hand and arm exercises. The MusicGlove is a glove that measures finger movements and allows its user to play a musical computer game using those movements. The RAE is a lever that attaches to a manual wheelchair with elastic bands and can be pushed back and forth to exercise the arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years of age
* Sustained a single stroke affecting the arm, at least three months prior to enrollment
* Minimal to moderate lost motor control of the arm after stroke
* No active major psychiatric problems, or neurological/orthopedic problems affecting the stroke-affected upper extremity
* No active major neurological disease other than the stroke
* Absence of pain in the stroke-affected upper extremity

Exclusion Criteria:

* Severe tone at the affected upper extremity
* Severe aphasia
* Severe reduced level of consciousness
* Severe sensory/proprioception deficit at the affected upper extremity
* Currently pregnant
* Difficulty in understanding or complying with instructions
* Inability to perform the experimental task that will be studied
* Increased pain with movement of the stroke-affected upper extremity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Cramer, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine, Irvine, California, United States

REFERENCES:
- [Derived] Zondervan DK, Friedman N, Chang E, Zhao X, Augsburger R, Reinkensmeyer DJ, Cramer SC. Home-based hand rehabilitation after chronic stroke: Randomized, controlled single-blind trial comparing the MusicGlove with a conventional exercise program. J Rehabil Res Dev. 2016;53(4):457-72. doi: 10.1682/JRRD.2015.04.0057. PMID 27532880
- [Derived] Zondervan DK, Augsburger R, Bodenhoefer B, Friedman N, Reinkensmeyer DJ, Cramer SC. Machine-Based, Self-guided Home Therapy for Individuals With Severe Arm Impairment After Stroke: A Randomized Controlled Trial. Neurorehabil Neural Repair. 2015 Jun;29(5):395-406. doi: 10.1177/1545968314550368. Epub 2014 Oct 1. PMID 25273359

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MusicGlove Group | Control Group for Music Glove | Resonating Arm Exerciser (RAE) | Control Group for RAE
Started | 11 | 12 | 9 | 8
Completed | 9 | 8 | 8 | 8
Not Completed | 2 | 4 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0 | 0
Not completed — unrelated injry | 1 | 1 | 0 | 0
Not completed — got a job | 0 | 1 | 0 | 0
Not completed — Got sick and could not complete study | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were 40 participants enrolled in the study, however 7 of them did not complete the study. We listed the 7 and their reasons of not completing study in section "participant flow overview".
Groups:
- Total: Total of all reporting groups
Arm/Group | MusicGlove Group | Control Group for Music Glove | Resonating Arm Exerciser (RAE) | Control Group for RAE | Total
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 33
Age, Continuous [Mean (Full Range); unit: years] | 60 [45 to 74] | 59 [35 to 74] | 61 [32 to 80] | 54 [39 to 76] | 60 [32 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 2 | 1 | 10
  Male | 5 | 5 | 6 | 7 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 8 | 7 | 7 | 7 | 29
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 6 | 4 | 5 | 4 | 19
  More than one race | 1 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 8 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Motor and Strength Outcome Measure Using Box and Block Test
Description: The primary end point was the change in Box and Blocks score, which measures how many blocks a subject can pick up and place in a box in 60 secons, from baseline to 1 month posttherapy. The higher the scores, the better arm and hand function indicated.
Time Frame: From baseline to 1 month post therapy
Population: Number of blocks participants able to pick up and place in a box in 60 seconds at one month follow up minus the number of blocks participants able to pick up and place in a box in 60 seconds at baseline. Please note that box and block test was the primary outcome measure for the Music Glove part of the study.
Measure: Mean (Standard Deviation); unit: blocks
Arm/Group | MusicGlove Group | Control Group for Music Glove
Number analyzed (Participants) | 9 | 8
blocks | 2.3 (6.2) | 4.3 (5.0)

2. Primary Outcome: Motor and Strength Outcome Measure Using Fugl-Meyer Score
Description: The primary outcome measure was the change in Upper Extremity FM score on a scale of 0 to 66 at one month post therapy. The higher the scores, the better arm and hand function indicated.
Time Frame: From baseline to 1 month post therapy
Population: Fugl-Meyer score at one month post therapy minus Fugl-Meyer score at baseline on a 66 point scale. Please note that Fugl-Meyer UE motor score is the primary outcome measure for RAE part of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Resonating Arm Exerciser (RAE) | Control Group for RAE
Number analyzed (Participants) | 8 | 8
units on a scale | 2.88 (4.68) | 1.31 (2.59)

3. Other Pre Specified Outcome: Range of Motion of Shoulder Joint
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | MusicGlove Group | Control Group for Music Glove | Resonating Arm Exerciser (RAE) | Control Group for RAE
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No